CLINICAL TRIAL: NCT04514978
Title: The Effect of Blood Donation on Hematological and Iron Indices and Detection of Autologous Blood Transfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: World Anti-Doping Agency (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nikolai Nordsborg, Associate professor, Head of Department, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H-17024876
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Blood Donation; Blood Transfusion

STUDY DESIGN:
Intervention Model Description: Explorative
Who Masked: Participant, Care Provider, Investigator
Masking Description: An algorithm was created using randomizer.org
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood donation and transfusion (Experimental): Donation and reinfusion of 1 unit whole blood and 130 mL packed red blood cells, respectively. Blood samples were collected at 8 weeks prior to donation for 12 subjects and 2 weeks prior to donation by 12 subjects. Blood samples were collected 3, 7, 14, 21, and 28 days after donation and 3, 6, 24 hours and 2, 3 and 6 days after reinfusion of blood.
  Interventions: Procedure: Blood donation and blood transfusion
- Control group (No Intervention): Blood samples collected with same frequency as described in the intervention arm.

INTERVENTIONS:
Procedure: Blood donation and blood transfusion — 24 subjects (12 female, 12 male) is phlebotomized and four weeks later ~130 mL packed red blood cells are re-infused in the same subjects.
  Arms: Blood donation and transfusion

SUMMARY:
Blood donations is a essential and crucial in the clinic. Normal biological variation of relevant biomarkers and hormones before the donation of 450 mL whole blood as well as the expected alterations in systemic levels of plasma iron indices and RBC measures up to 4 weeks after donation in healthy, non-anemic, young men and women is investigated

Likewise, the possibilities for detecting autologous blood transfusion is investigated.

DETAILED DESCRIPTION:
Blood donations is a essential and crucial in the clinic. A whole blood donation results in the loss of 450-525 mL whole blood in eight to ten minutes and is known to reduce body iron stores with 200-265 mg iron depending on the donor's age, hematocrit and sex and accounts for 25% of average tissue iron stores in men and up to 75% in women.In the present study, the investigators aimed at thoroughly evaluate normal biological variation of relevant biomarkers and hormones before the donation of 450 mL whole blood as well as the expected alterations in systemic levels of plasma iron indices and red blood cell measures up to 4 weeks after donation in healthy, non-anemic, young men and women

Likewise, doping in sport is a major problem concerning both the health of the athletes and the integrity of sports. Despite major improvements in anti-doping work in recent years, it is still impossible to test for all existing and future doping strategies, such as manipulation with blood oxygen carrying capacity. A well-known doping strategy is autologous blood transfusion (ABT), and at present, the detection of ABT is a challenge for anti-doping authorities. The hypotheses for this study are that 1) ret% and abnormal blood profile score (ABPS) have higher sensitivity to micro-dose ABT compared to current variables in the Athlete Biological Passport (ABP); 2) The plasma concentration of hepcidin and erythroferrone (ERFE) is sensitive to micro-dose ABT; 3) Gender-specific variations in hematologic variables affect the interpretation of the athlete's biological passport.

ELIGIBILITY:
Inclusion Criteria:

* Relative maximum oxygen uptake (VO2-max) of at least 55 ml O2/min/kg for male participants and 50 ml O2/min/kg for female participants

Exclusion Criteria:

* Age
* Insufficient fitness level
* Blood donation 3 months prior to enrollment
* Altitude exposure 2 months before enrollment
* Hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin centration | 6 days after reinfusion
  The effect of the intervention on [Hb] levels will be investigated
reticulocyte percentage | 6 days after reinfusion
  The effect of the intervention on ret% levels will be investigated
OFF-score | 6 days after reinfusion
  The effect of the intervention on OFF-score (an algorithm computed from reticulocyte percentage and hemoglobin concentration resulting in a arbitrary value) will be investigated
Homeostatic markers of iron metabolism | 6 days after reinfusion
  Markers of iron metabolism such as hepcidin and erythroferrone are collected and analyzed for evaluation of iron metabolism during and after donation and reinfusion of blood.

SECONDARY OUTCOMES:
Endurance exercise performance measured as a preloaded 400 kcal time-trial | 6 days after reinfusion.
  Endurance exercise performance are measured in a subgroup of 13 subjects.
Maximal oxugen uptake (VO2max) | 6 days after reinfusion.
  Maximal aerobic capacity is measured via a maximal oxygen uptake incremental test in a subgroup of 13 subjects.
Mean corpuscular concentration | 6 days after reinfusion.
  Markers of red blood cell size and hemoglobin content are collected and analyzed for Determining the impact of donation and reinfusion of blood.
Mean corpuscular hemoglobin concentration | 6 days after reinfusion.
  Markers of red blood cell size and hemoglobin content are collected and analyzed for Determining the impact of donation and reinfusion of blood.
Mean corpuscular volume | 6 days after reinfusion.
  Markers of red blood cell size and hemoglobin content are collected and analyzed for Determining the impact of donation and reinfusion of blood.
Dried Blood Spots | 6 days after reinfusion.
  Dried blood spots will be analyzed for the CD71/Band3 concentration as well as transcriptomic markers for reticolucytes including the ALAS2 L and LC.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymous data will be shared with other researchers.

REFERENCES:
- [Derived] Breenfeldt Andersen A, Bejder J, Bonne TC, Sorensen H, Sorensen H, Jung G, Ganz T, Nemeth E, Secher NH, Johansson PI, Nordsborg NB. Hepcidin and Erythroferrone Complement the Athlete Biological Passport in the Detection of Autologous Blood Transfusion. Med Sci Sports Exerc. 2022 Sep 1;54(9):1604-1616. doi: 10.1249/MSS.0000000000002950. Epub 2022 Apr 25. PMID 35482790